CLINICAL TRIAL: NCT03387592
Title: A Randomized Phase II Trial of Capecitabine and Temozolomide (CAPTEM) or FOLFIRI as SEcond-line Therapy in NEuroendocrine CArcinomas and Exploratory Analysis of Predictive Role of Positron Emission Tomography (PET) Imaging and Biological Markers
Brief Title: CAPTEM or FOLFIRI as SEcond-line Therapy in NEuroendocrine CArcinomas
Acronym: SENECA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efficacy endpoint not met according to first step of Briant-Day design
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST100.22
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2022-03

CONDITIONS: Neuroendocrine Carcinoma
Keywords: Neuroendocrine Carcinoma; second line therapy; PET imaging; FOLFIRI; CAPTEM
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Irinotecan; Fluorouracil; Capecitabine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFIRI regimen (Active Comparator): CPT-11 180 mg/m2, given as 60 min. i.v. infusion on day 1 every 2 weeks followed by Calcio levofolinate 200 mg/m2, given as a 2h i.v. infusion on days 1 every 2 weeks followed by 5-Fluorouracil 400 mg/m2 given as bolus, and then 5-Fluorouracil 2400 mg/m2 given as a 48 h continuous infusion on day 1, every 2 weeks, until progression or for a maximum of 12 cycles
  Interventions: Drug: CPT-11; Drug: Calcio levofolinate; Drug: 5-Fluorouracil
- CAPTEM regimen (Experimental): Capecitabine 750 mg/m2 twice a day on days 1-14 in combination with Temozolomide 200 mg/m2 daily on days 10-14, every 4 weeks, until progression or for a maximum of 6 cycles
  Interventions: Drug: Capecitabine; Drug: Temozolomide

INTERVENTIONS:
Drug: CPT-11 — 180 mg/m2
  Arms: FOLFIRI regimen
Drug: Calcio levofolinate — 200 mg/m2
  Arms: FOLFIRI regimen
Drug: 5-Fluorouracil — 400 mg/m2 + 2400 mg/m2
  Arms: FOLFIRI regimen
Drug: Capecitabine — 1500 mg/m2
  Arms: CAPTEM regimen
Drug: Temozolomide — 200 mg/m2
  Arms: CAPTEM regimen

SUMMARY:
This is a randomized phase II non comparative study. Patients with metastatic Neuroendocrine Carcinomas (NEC) Grade 3, will be enrolled in the study and will be randomly assigned to receive FOLFIRI or CAPTEM as second line treatment. Disease control rate (DCR) and safety are primary objectives, secondary objectives are Disease control rate (OS), Progression Free Survival (PFS), quality of life and toxicity of subsequent line of therapy (after Progression Disease PD) with an observational purpose.

DETAILED DESCRIPTION:
This is a multicenter randomized phase II non comparative study. Patients with metastatic NEC G3, will be enrolled in the study and will be randomly assigned to receive FOLFIRI or CAPTEM as second line treatment The primary objective is to assess DCR and the safety as co-primary objective. The secondary objectives are: OS, PFS, quality of life and toxicity of subsequent line of therapy (after Progression Disease PD) with an observational purpose.

The secondary exploratory objectives are the assessment of the impact of PET with gallium on PFS and the evaluation of biomarkers

Study treatment:

FOLFIRI regimen

* Oxaliplatin (CPT-11) 180 mg/m2, given as 60 min. i.v. infusion on day 1 every 2 weeks followed by
* Calcio levofolinate 200 mg/m2, given as a 2h i.v. infusion on days 1 every 2 weeks followed by
* 5-Fluorouracil 400 mg/m2 given as bolus, and then 5-Fluorouracil 2400 mg/m2 given as a 48 h continuous infusion on day 1, every 2 weeks, until progression or for a maximum of 12 cycles

CAPTEM regimen Capecitabine 750 mg/m2 twice a day on days 1-14 in combination with temozolomide 200 mg/m2 daily on days 10-14, every 4 weeks, until progression or for a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologic diagnosis of neuroendocrine carcinomas (GEP NEC and lung NEC), G3 with ki67 > 20%. Other rare sites of origin such as genitourinary or gynecological or larynx or unknown origin neuroendocrine carcinoma with Ki67 > 20% will be included.
2. Male or Female, aged >=18 years.
3. Measurable disease according to RECIST 1.1 criteria.
4. Patients who already received a first line treatment for metastatic disease with platinum compound-based regimen chemotherapy (Cisplatin/Carboplatin and Etoposide, folfox4 or Capecitabine-Oxaliplatin).
5. Previous treatments with immuno checkpoint-inhibitor and/or everolimus are permitted
6. Life expectancy greater than 3 months
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
8. Adequate haematological, liver and renal function:

   neutrophils > 2.0 x 109 /L, platelet > 100 x 109 /L, hemoglobin > 10g/dL, total bilirubin < 1 Upper Normal Limit (UNL), Aspartate aminotransferase (ASAT) and Alanine transaminase (ALAT) < 2.5 x UNL or < 5 x UNL in presence of liver metastases, alkaline phosphatase < 2.5 x UNL; patients with ASAT or ALAT >1.5 x UNL associated with alkaline phosphatase >2.5 x UNL are not eligible.); creatinine <1.5 UNL. In presence of borderline values, the calculated creatinine clearance according to Cockcroft-Gault formula, 60 ML/min.
9. If female of childbearing potential highly effective birth control methods, according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials", (2014_09_15 section 4.1) are mandatory. Highly effective birth control methods are required beginning at the screening visit and continuing until 6 months following last treatment with study drug. Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 6 months after final study drug administration. Two acceptable methods of birth control thus include Condom (barrier method of contraception) and one of the following is required ( established use of oral, or injected or implanted hormonal method of contraception by the female partner; placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner; additional barrier method like occlusive cap with spermicidal foam/gel/film/cream/suppository in the female partner; tubal ligation in the female partner; vasectomy or other procedure resulting in infertility (eg, bilateral orchiectomy), for more than 6 months.
10. Written informed consent signed and dated before registration procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirement.
11. Brain metastases allowed if asymptomatic at study baseline. Whole brain irradiation or focal treatment for Central Nervous System (CNS) metastases are permitted.

Exclusion Criteria:

1. Ki67 index ≤ 20 %.
2. Patients with metastatic NECs already treated with irinotecan regimen.
3. Patients with a known hypersensitivity to fluorouracil or calcium levofolinate or Irinotecan or their recipients.
4. All acute toxic effects of any prior therapy (including surgery radiation therapy, chemotherapy) must have resolved to a grade <= 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE).
5. Life expectancy minor than 3 months.
6. ECOG performance status >2.
7. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
8. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

   * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
   * severely impaired lung function (spirometry and diffusing capacity of lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or Oxygen saturation that is 88% or less at rest, in room air).
   * uncontrolled diabetes as defined by fasting serum glucose >1.5 x UNL.
   * any active (acute or chronic) or uncontrolled infections/disorders
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition.
10. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
11. Patients with uncontrolled or symptomatic brain metastases will be excluded because they often develop progressive neurologic dysfunction that can be confounding of neurologic and other adverse events
12. Other malignancy with a disease-free interval of less than 5 years (except non melanoma skin cancer or low grade superficial bladder cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | responses to treatment lasting at least 12 weeks up to 48 months of study period
  DCR is defined as the percentage of patients who have achieved complete, partial response and stable disease lasting for at least 12 weeks. DCR will be evaluated using the new international criteria proposed by the Version 1.1 Response Evaluation Criteria in Solid Tumors (RECIST).
Incidence of treatment related adverse events | up to 60 months
  Acute treatment related adverse events and late treatment related adverse events will be evaluated; the late treatment related adverse events is the adverse event that occurred after 30 days from the last treatment cycle. The adverse events will be evaluated according to CTCAE Version 5.0.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 60 months
  Overall Survival (OS) is defined as the time from treatment start to the time of death from any cause. Subjects who are alive at the time of the final analysis or who have become lost to follow-up will be censored at their last known alive date.
Progression Free Survival (PFS) | up to 60 months
  Progression free survival is defined as the time from the start treatment date to the date of first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.
Objective response rate (ORR) | responses to treatment lasting at least 12 weeks up to 60 months of study period
  ORR is defined as the percentage of patients who have achieved complete and partial response for at least 12 weeks from therapy start.
Quality of Life Questionnaire (QLQ) | up to 60 months
  Quality of life will be evaluated through validated standardized data collection forms from the EORTC QLQ-C30 questionnaire (quality of life questionnaire). Scoring of global health status, functional scales and symptom scales will be calculated according to EORTC QLQ-C30 Scoring Manual.
Evaluation of biomarkers | up to 60 months
  testing for mutational status of Multiple endocrine neoplasia, type 1 (MEN1), death-domain-associated protein (DAXX), α thalassemia/mental retardation syndrome X-linked (ATRX) and Retinoblastoma 1 (RB-1) on primary tumors tissues and for miRNA on blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Toni Ibrahim, MD, Principal Investigator — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)
Locations (23):
- Italy (23):
  - Az. Osp. Ospedali Riuniti di Ancona, Ancona, AN
  - A.O.U. Policlinico di Bari, Bari, BA
  - IRCCS IST. Tumori Bari - Giovanni Paolo II, Bari, BA
  - Ospedale di Feltre, Feltre, Belluno
  - ASST Spedali Civili di Brescia, Brescia, BS
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC
  - AOU Careggi, Florence, FI
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Nazionale Tumori Milano, Milan, MI
  - Azienda Ospedaliera-Universitaria di Modena, Modena, MO
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone", Palermo, PA
  - Centro di Riferimento Oncologico di Aviano, Aviano, Pordenone
  - Ospedale Civile degli Infermi, Faenza, RA
  - Policlinico Campus Biomedico Roma, Roma, RM
  - AOU San Luigi Gonzaga, Orbassano, TO
  - Azienda Ospedaliere Universitaria Integrata Verona, Verona, VR
  - Policlinico S. Orsola-Malpighi, Bologna
  - Ospedale di Bolzano, Bolzano
  - IRCCS "Saverio De Bellis", Castellana Grotte
  - Ospedale "Vito Fazzi", Lecce
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera-Universitaria di Parma, Parma
  - Ospedale S.Chiara - AOU Pisana, Pisa

REFERENCES:
- [Derived] Bongiovanni A, Liverani C, Foca F, Bergamo F, Leo S, Pusceddu S, Gelsomino F, Brizzi MP, Di Meglio G, Spada F, Tamberi S, Lolli I, Cives M, Marconcini R, Pucci F, Berardi R, Antonuzzo L, Badalamenti G, Santini D, Recine F, Vanni S, Tebaldi M, Severi S, Rudnas B, Nanni O, Ranallo N, Crudi L, Calabro L, Ibrahim T. A randomized phase II trial of Captem or Folfiri as second-line therapy in neuroendocrine carcinomas. Eur J Cancer. 2024 Sep;208:114129. doi: 10.1016/j.ejca.2024.114129. Epub 2024 May 25. PMID 39002347
- [Derived] Bongiovanni A, Liverani C, Pusceddu S, Leo S, Di Meglio G, Tamberi S, Santini D, Gelsomino F, Pucci F, Berardi R, Lolli I, Bergamo F, Ricci S, Foca F, Severi S, Ibrahim T; SENECA Study Team Investigators. Randomised phase II trial of CAPTEM or FOLFIRI as SEcond-line therapy in NEuroendocrine CArcinomas and exploratory analysis of predictive role of PET/CT imaging and biological markers (SENECA trial): a study protocol. BMJ Open. 2020 Jul 19;10(7):e034393. doi: 10.1136/bmjopen-2019-034393. PMID 32690499